CLINICAL TRIAL: NCT06766162
Title: Virtual Reality and Endoscopic Mucosal and Submucosal Dissection: a Patient Centred Experience "VREMRESD"
Brief Title: Virtual Reality to Improve Patient Experience During Endoscopic Mucosal and Submucosal Resection
Acronym: VREMRESD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24/LO/0785; 345381 (Other: IRAS)
Record Dates: First submitted 2024-12-16; First posted 2025-01-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: VR; Virtual Reality Pain Distraction; Endoscopic Submucosal Dissection; Endoscopic Mucosal Resection
Keywords: VRESD; Virtual reality and ESD; VR and endoscopic submucosal dissection; Virtual reeality and endoscopic submucosal dissection; VRWMR; VREMRESD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) Arm (Experimental): The VR arm will have a trial run with the VR headset in the endoscopy admission unit. The VR will then be applied at the start of the procedure. If, during the procedure, the patient requests sedation or pain medication, it will be provided. If the patient wishes to remove the VR headset, they may do so at any time.
  Interventions: Other: Virtual reality pain distraction
- Standard Arm (Active Comparator): The control group will follow the standard local protocol for analgesia and sedation throughout the procedure.
  Interventions: Other: Standard analgesia and sedation

INTERVENTIONS:
Other: Virtual reality pain distraction — The intervention group in this study will undergo their EMR and ESD procedure with the addition of virtual reality (VR) as a supportive tool. Participants in this group will use a VR headset during the procedure, designed to provide an immersive experience that may help manage pain and anxiety. The use of VR will be integrated alongside the standard care protocol, including routine sedation and pain management practices VR headset is from DRVR, Rescope innovation which is registered as medical device in the UK.
  Arms: Virtual reality (VR) Arm
Other: Standard analgesia and sedation — Standard local protocol for analgesia and sedation, incorporating fentanyl and midazolam.
  Arms: Standard Arm

SUMMARY:
This study explores the feasibility of using Virtual Reality (VR) to manage pain and anxiety during Endoscopic Mucosal (EMR) and Submucosal Dissection (ESD). EMR and ESD often requires sedation or analgesia, which can cause side effects like respiratory or cardiac suppression. VR, by immersing patients in a calming virtual environment, has shown potential in reducing pain and anxiety in medical settings. This study aims to evaluate its application in improving pain management and reducing sedation use during EMR and ESD.

DETAILED DESCRIPTION:
This study utilizes a prospective randomized controlled trial (RCT) design to evaluate the feasibility of incorporating Virtual Reality (VR) as a method for pain management during Endoscopic mucosal and (EMR) Submucosal Dissection (ESD). Participants will be randomized into two groups: one receiving VR sedation with on-demand analgesia and sedation, and the other following standard sedation protocols. The primary endpoint is to assess the feasibility of integrating VR for pain management during EMR or ESD procedures.

Eligibility criteria ensure that participants are suitable for the study. Patients must be 18 years or older, scheduled for EMR ESD, able to provide informed consent, and proficient in English. Those with contraindications for EMR, ESD, severe impairments affecting VR use, or conditions contraindicating VR are excluded. Endoscopists must be experienced in EMR and ESD, willing to participate, and fluent in English, with non-ESD practitioners or those unwilling to participate excluded.

The study aims to enroll 40 patients (20 per group) and involve five experienced endoscopists from the unit, all of whom will be consented. Secondary endpoints include the proportion of EMR and ESD procedures completed using VR, reductions in sedation and analgesia usage, differences in pain scores between the two groups, and satisfaction levels of both patients and endoscopists.

Follow-up will consist of immediate post-procedure feedback and questionnaires to gather insights on VR's impact. This trial will provide critical data on the potential for VR to enhance patient experience, optimize sedation use, and improve procedural outcomes during EMR and ESD, informing future research and clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to consent.
* Fit to use virtual reality.
* Patients allocated to appropriate EMR/ ESD lists.

Exclusion Criteria:

* Patients who are unable to consent.
* Contraindication to use VR including, epilepsy and photosensitivity.
* Planned other interventional colonoscopy (Polypectomy, Stenting).
* Visually impaired.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility for integrating VR as a pain mediation during EMR/ESD procedure. | During the EMR/ESD procedure
  This will evaluteed by:
  The completed numbers of ESD procedure with the use of the VR as an additive measure to recduce the need for analgesia and sedation.

SECONDARY OUTCOMES:
The change in analgesia and sedation used while using the VR. | During the EMR/ESD prcoedure
  This will be evaluated by calculating the mean amount of diazepam and fentanyl used in both groups to compare the standard pathway for analgesia and sedation with the VR intervention.
The difference in pain scores between the two groups. | baseline, pre-procedure, immediately after the procedure
  Pain scores will be evaluated by collecting pain scores on a Likert scale from 0 to 10, where 0 means no pain and 10 indicates maximum pain. The mean values will be compared between the two groups.
Patient satisfaction. | immediately after the procedure
  Patient satisfaction will be evaluated by collecting satisfaction scores on a Likert scale from 0 to 10, where 0 means completely dissatisfied and 10 indicates completely satisfied. The mean values will be compared between the two groups.
Endoscopist satisfaction. | immediately after the procedure
  Endoscopist satisfaction with performing EMR/ESD using VR or standard intervention groups will be evaluated by collecting satisfaction scores on a Likert scale from 0 to 10, where 0 means completely dissatisfied and 10 indicates completely satisfied. The mean values will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- king's College Hospitals, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Q, Zang Y, Zang W, Cai W, Li W, Guo Y, Xin C, Tu X. Implementation of virtual reality technology to decrease patients' pain and nervousness during colonoscopies: a prospective randomised controlled single-blinded trial. Clin Med (Lond). 2022 May;22(3):237-240. doi: 10.7861/clinmed.2022-0001. Epub 2022 Apr 20. PMID 35443967
- [Background] Karaveli Cakir S, Evirgen S. The Effect of Virtual Reality on Pain and Anxiety During Colonoscopy: A Randomized Controlled Trial. Turk J Gastroenterol. 2021 May;32(5):451-457. doi: 10.5152/tjg.2021.191081. PMID 34231475